CLINICAL TRIAL: NCT05805579
Title: Prognostic Value of Transthoracic Diaphragmatic Echography in COVID-19 Pneumonia Patients With Acute Respiratory Failure
Brief Title: Diaphragmatic Echography in COVID-19 Pneumonia
Acronym: COVIDUSDIAP
Status: Completed | Type: Observational
Sponsor: Javier Lázaro (Other)
Collaborators: Sociedad Aragonesa de Patología del Aparato Respiratorio (Unknown)
Responsible Party: Sponsor-Investigator, Javier Lázaro, MD; PhD, Aragon Institute of Health Sciences
Organization: Aragon Institute of Health Sciences (Other)
Other Study IDs: ROYO1
Record Dates: First submitted 2023-04-03; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Pneumonia, Viral; Covid19; Respiratory Failure
Keywords: COVID19 pneumonia; Diaphragm ultrasound
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diaphragmatic echography — Diaphragmatic echography

SUMMARY:
We hypothesized that diaphragm thickness is concerned in acute respiratory failure of COVID19 patients and its ultrasound measure at the begining of hospitalisation is a good predictor of poor outcome.

A prospective observational non intervention study is designed.

DETAILED DESCRIPTION:
To answer our hypothesis we will perform diaphragm ultrasound in the first 24hr hospitalized COVID19 patients.

In the ultrasound exploration we will assess diaphragm movility and thickness. We will also assess other clinical, biochemistry and radiological variables. The main outcome we want to analyze is the destination on discharge: home, respiratory intermediate critical unit or exitus.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 Pneumonia Acute respiratory failure (PaO2 <60mmHg)

Exclusion Criteria:

* Invasive or non invasive ventilation within first 24h Neuromuscular disease Diaphragmatic paralysis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People hospitalaised in pulmonology service
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Early diaphragm ultrasound as a predictor factor for invasive and non invasive ventilation and death | From date of inclusion until discharge date (lenght of hospitalization)
  This is the main outcome of our study given that it has a important clinical implications. If we confirm our hypothesis diaphragm ultrasound could prove to be a useful prognosis tool for COVID19 patients.

SECONDARY OUTCOMES:
Diaphragm thickness rate as a predictor factor for invasive and non invasive ventilation and death | From date of inclusion until discharge date (lenght of hospitalization)
  Diaphragm strenght is directly related to thickness. The impact of COVID19 infection on this specific measure can predict patient evolution.
Diaphragm movility rate as a predictor factor for invasive and non invasive ventilation and death | From date of inclusion until discharge date (lenght of hospitalization)
  Diaphragm fatigability is directly related to movility. The impact of COVID19 infection on this specific measure can predict patient evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Javier Lázaro Sierra, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
All investigators that can use these data are included as collaborators. Sharing that type of information is forbiden by our ethics comitee

REFERENCES:
- [Background] Marchioni A, Castaniere I, Tonelli R, Fantini R, Fontana M, Tabbi L, Viani A, Giaroni F, Ruggieri V, Cerri S, Clini E. Ultrasound-assessed diaphragmatic impairment is a predictor of outcomes in patients with acute exacerbation of chronic obstructive pulmonary disease undergoing noninvasive ventilation. Crit Care. 2018 Apr 27;22(1):109. doi: 10.1186/s13054-018-2033-x. PMID 29703214
- [Background] Pivetta E, Cara I, Paglietta G, Scategni V, Labarile G, Tizzani M, Porrino G, Locatelli S, Calzolari G, Morello F, Maule MM, Lupia E. Diaphragmatic Point-of-Care Ultrasound in COVID-19 Patients in the Emergency Department-A Proof-of-Concept Study. J Clin Med. 2021 Nov 14;10(22):5291. doi: 10.3390/jcm10225291. PMID 34830573
- [Background] Schepens T, Fard S, Goligher EC. Assessing Diaphragmatic Function. Respir Care. 2020 Jun;65(6):807-819. doi: 10.4187/respcare.07410. PMID 32457172
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Derived] Lazaro Sierra J, Doz Arcas M, Claveria Marco P, Rosell Abos MT, Santolaria Lopez MA, Perez Gimenez L, Lanzuela Benedicto T, Zuil Martin M, Boldova Loscertales A, Garcia Saez S, Huertas Puyuelo A, Nieto Sanchez D, Carretero Garcia JA. Prognostic Value of Diaphragmatic Ultrasound in Patients Admitted for COVID-19 Pneumonia. Open Respir Arch. 2023 Dec 1;6(1):100290. doi: 10.1016/j.opresp.2023.100290. eCollection 2024 Jan-Mar. PMID 38293643